CLINICAL TRIAL: NCT01250262
Title: Resistance Exercise Effects on Fear Avoidance Beliefs and Physical Function in Obese, Older Adults With Chronic Low Back Pain
Brief Title: Resistance Exercise Effects on Fear Avoidance and Physical Function in Obese Older Adults With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 258-2010
Record Dates: First submitted 2010-11-05; First posted 2010-11-30 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Low Back Pain; Obesity
Keywords: low back pain; obese; fear avoidance; disability and low back pain; chronic low back pain in obese older adults
MeSH Terms: conditions — Low Back Pain; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard care (Active Comparator): Subjects will receive normal medical care and follow up during the four month study period if assigned to this group.
  Interventions: Other: normal medical care and follow up
- Isolated Lumbar Resistance Exercise Program (Active Comparator): Lumbar extension exercise protocol to increase strength and reduce pain.
  Interventions: Other: Isolated Lumbar Resistance Exercise Program
- Total Body Resistance Exercise Program (Active Comparator): Training protocol for 1 set for each exercise: leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, calf press and abdominal curl
  Interventions: Other: Total Body Resistance Exercise Program

INTERVENTIONS:
Other: normal medical care and follow up — physical activity/ nutrition guidelines will be provided and reviewed with the participant as part of standard care; telephone contact will be made weekly to encourage adherence to the health guidelines
  Arms: Standard care
Other: Isolated Lumbar Resistance Exercise Program — lumbar extension, two set of 10-15 repetitions, once a week for two weeks; lumbar extension, one set of 10-15 repetitions, three times a week, week 3 to 4 months
  Arms: Isolated Lumbar Resistance Exercise Program
Other: Total Body Resistance Exercise Program — exercises: leg press, leg curl, leg extension, chest press, seated row, overhead press, triceps dip, biceps curl, calf press and abdominal curl, one set of 10-12 repetitions, three time per week, week one to 4 months
  Arms: Total Body Resistance Exercise Program

SUMMARY:
The purpose of this study is to determine if a 4 month resistance exercise program reduces the severity of low back pain, pain-related fear avoidance and improves mobility compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain for >6 months
* >3 pain episodes per week
* waist circumferences ≥102 cm for men
* waist circumferences ≥ 88 cm for women
* willing and able to participate in regular exercise for 14 weeks
* using pain medications to control low back pain
* free of abnormal cardiovascular responses during a screening graded maximal walk test

Exclusion Criteria:

* unable to walk
* participating in regular resistance exercise training (>3X week) in the past 6 months
* pain symptoms are too severe and prevent strength testing or walking
* acute back injury
* spinal stenosis that precludes walking one block due to neurogenic claudication
* back surgery within the past 2 years
* current use of weight loss interventions (drugs; exercise interventions)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
10 centimeter Visual Analog Scale (VAS); Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3 and 4 Months
  The VAS scale will range from 0-10 cm, where a rating of "0" reflects no pain, and a "10" rating represents "worst pain imaginable. Subjects will complete the VAS at the indicated time intervals to document any change in their pain levels.
Tampa Scale of Kinesiophobia (TSK); Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3 and 4 Months
  Fear avoidance beliefs will be measured using the 11 item TSK. Subjects will complete the TSK at the indicated time intervals to document any change in their fear avoidance beliefs.
Fear-Avoidance Beliefs Questionnaire (FABQ); Change from Baseline at 1, 2, 3 and 4 Months | Baselinje, 1, 2, 3 and 4 Months
  The FABQ is a tool based on theories of fear and avoidance behavior and focuses specifically on beliefs about how physical activity and work affect low back pain. Subjects will complete the FABQ at the indicated time intervals to document any change in their fear and avoidance behavior.
Pain Catastrophizing Scale (PCS); Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3 and 4 Months
  The PCS will be used to assess the effect of the chronic back pain on rumination on pain symptoms and helplessness. Subjects will complete the PCS at the indicated time intervals to document any change in their thoughts of their pain symptoms.
Modified Oswestry Disability Index (ODI); Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3 and 4 Months
  The ODI is responsive to intervention treatments for low back pain, is reliable, and corresponds well with several global patient disability measures. Subjects will complete the ODI at the indicated time intervals to document any change in their low back pain.
Roland Disability Survey (RDS); Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3, and 4 Months
  The RDS assesses physical disability and mental function with low back pain; this survey is sensitive to treatment interventions, and is reproducible and consistent and correlated well with other global ratings and disability measures. Subjects will complete the RDS at the indicated time intervals to document any change in their physical disability and mental function with their low back pain.

SECONDARY OUTCOMES:
Graded Treadmill Exercise Test; Change from Baseline at 4 Months | Baseline and 4 Months
  Maximal aerobic fitness, or oxygen consumption (VO2max) will be determined using a walking symptom-limited graded exercise test. Subjects will complete the exercise test at the indicated time intervals to document any change in their aerobic fitness.
Chair Rise Time, Stair Climb Time and Gait Assessment; Change from Baseline at 4 Months | Baseline and 4 Months
  Chair rise time will be measured as the participant moves from a sitting to a full standing position. The time to walk up one flight of stairs will be measured by having the participants walk up one flight of stairs consisting of 12 steps as quickly as possible. Gait will be assessed by having the participants walk across a 26' portable walkway. Subjects will complete these motions at the indicated time intervals to document any change.
7-day Pedometer Test; Change from Baseline at 4 Months | 7 day period at Baseline and 4 Months
  Community ambulation will be estimated using a 7-day pedometer test in which participants will wear a StepWatch® step activity monitor. Subjects will complete this test at the indicated time intervals to document any change in their ambulation.
Ultrasound Muscle Thickness; Change from Baseline at 4 Months | Baseline and 4 Months
  The ultrasound technique that will be used to capture muscle thickness changes in the paraspinal and multifidus muscles. Subjects will be tested at the indicated time intervals to document any change.
Muscle Strength; Change from Baseline at 1, 2, 3 and 4 Months | Baseline, 1, 2, 3 and 4 Months
  Assessments of strength (1 repetition maximum, 1-RM) will be determined for all muscle groups trained. Subjects will be assessed at the indicated time intervals to document any change.

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Vincent, Ph.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States